CLINICAL TRIAL: NCT04197102
Title: Use of Cannabidiol (CBD) Oil in the Treatment of PTSD: A Placebo-Controlled Randomized Clinical Trial
Brief Title: Use of CBD Oil in the Treatment of Posttraumatic Stress Disorder
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Suspended (The UT IRB determined that CBD oil is being used as a drug as defined by the FDA. Therefore, an IND must be obtained for the use of CBD oil in this research study in accordance with FDA regulations, 21 CFR 312.)
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Professor of Psychology, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-05-0123
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD, CBD, cannabidiol, home-based study
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Color Vision Defects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each nightly dose of CBD/Placebo oil will be tagged with a code # on the plastic syringe containing the CBD oil or placebo oil. All oils will have identical color and mint flavor. Two independent staff not connected to the study will be unblinded to the participants' assignment to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBD Isolate (Active Comparator): 300 mg/day of CBD isolate
  Interventions: Drug: CBD Isolate
- CBD Broad Spectrum (Active Comparator): 300 mg/day of CBD Broad Spectrum Oil
  Interventions: Other: CBD Broad Spectrum
- Placebo oil (Placebo Comparator): Matched Placebo Oil
  Interventions: Other: Placebo oil

INTERVENTIONS:
Drug: CBD Isolate — A fixed dose of 300-mg of a hemp-derived formulation of purified 99.9% CBD isolate oil will be taken once daily for 8 weeks for participants randomized to the CBD Isolate arm.
  Other Names: CBD Isolate Oil
  Arms: CBD Isolate
Other: CBD Broad Spectrum — A fixed dose of 300-mg of a hemp-derived formulation of purified 99.9% CBD Broad Spectrum oil will be taken once daily for 8 weeks for participants randomized to the CBD - Broad Spectrum arm.
  Other Names: CBD Broad Spectrum Oil
  Arms: CBD Broad Spectrum
Other: Placebo oil — Placebo solution will be taken once daily for 8 weeks by participants randomized to the placebo arm.
  Other Names: PLBO
  Arms: Placebo oil

SUMMARY:
The overarching objective of the proposed project is to test the clinical efficacy of CBD in the treatment of post-traumatic stress disorder using a rigorous double-blind randomized clinical trial methodology. Participants (n=150) meeting full DSM-5 criteria for post-traumatic stress disorder (PTSD) will be randomized to one of 3 treatment arms: (a) CBD -Isolate; (b) CBD-Broad Spectrum; (c) Placebo oil.

We predict that patients receiving CBD isolate or CBD Broad Spectrum will show significantly greater improvements in PTSD symptoms and functional impairment at the posttreatment and one-month follow-up relative to patients receiving placebo oil. Additionally, we expect that patients receiving CBD Broad Spectrum will show significantly greater improvements relative to patients receiving CBD Isolate.

DETAILED DESCRIPTION:
Background and Significance of the Proposed Project

Over 80% of Americans are exposed to a significant trauma sometime during their lifetime and approximately 7% will meet for a threshold diagnosis of posttraumatic stress disorder. PTSD is the most costly anxiety-related disorder and confers significant interference in work, social functioning, increased risk for other physical and mental health problems, and a four-fold increase in suicide rates compared to the general population.

Over the past two decades, trauma-focused psychotherapies for PTSD have been shown to outperform more traditional supportive psychotherapy or pharmacotherapy and have become the first line treatment for PTSD. Despite these advances, trauma focused treatments such as prolonged exposure therapy (PE) are associated with high rates of treatment refusal, and among those who do enter treatment, approximately 25% drop-out. These data highlight the need to develop PTSD treatment strategies that are both effective and more palatable to patients.

More recently, there's been considerable excitement in the press over the potential therapeutic use of cannabidiol (CBD) products in the treatment of a variety of physical and mental health problems.( Delta-9-tetrahydrocannabinol (delta-9 THC) is still illegal in most states because of its psychoactive abuse potential. In contrast, cannabidiol (CBD) does not convert to THC in the body and has negligible side effects relative to main stream psychiatric drugs (benzodiazepines and antidepressants) commonly prescribed for the treatment of PTSD. Mounting evidence from studies with rodents suggests that CBD may confer significant promising health-related benefits including anti-inflammatory, pain-relieving, anti-cancer, memory enhancement, and facilitation of fear extinction (see White for a recent review).

The biggest success story for CBD use in humans to date comes from controlled randomized clinical trials demonstrating a 50% or more reduction in previously intractable seizures in children suffering from Dravet syndrome and Lennox-Gastaut syndrome. Moreover, several controlled clinical trials have shown promising findings in reducing psychotic symptoms among patients with schizophrenia and among young adults displaying THC-induced psychosis.

Preliminary Evidence that CBD may offer promise in the treatment of anxiety-related disorders has started to emerge. A small pilot trial with 24 patients presenting with social anxiety disorder found that relative to placebo, a single dose of 100 mg of CBD oil led to lower levels of anxiety, cognitive impairment, and discomfort in their actual speech performance as well as their anxiety before the speech. Unfortunately, human treatment studies for anxiety-related problems is limited almost exclusively to single dose effects on an anxiety challenge task. Studies are clearly needed to assess the effects of multi-dose CBD treatments across the full spectrum of trauma and anxiety-related disorders such as posttraumatic stress disorder.

PROJECT AIMS

The overarching objective of the proposed project is to test the clinical efficacy of CBD in the treatment of posttraumatic stress disorder using a rigorous double-blind randomized clinical trial methodology.

Specific aims of the project include:

1. Compare the efficacy of an 8-week multi-dose regimen of two CBD oil formulations (CBD Isolate (300 mg/day) and CBD Broad Spectrum) relative to placebo oil in reducing PTSD symptoms at the posttreatment and one-month follow-up.

   We predict that patients receiving CBD oil (CBD isolate or CBD Broad Spectrum) will show significantly greater improvement in PTSD symptoms and functional impairment at post-treatment and one-month follow-up relative to patients receiving placebo oil.

   We also predict that patients receiving the CBD Broad Spectrum formulation will show significantly greater improvement in PTSD symptoms and functional impairment relative to patients receiving CBD Isolate.
2. Examine predictors of patients' clinical response to the various treatment combinations.

   We expect that the superiority of CBD relative to placebo will be more pronounced for patients showing more severe PTSD symptoms at baseline.
3. Examine the perceived acceptability and patients' side effects profile of 8 weeks of daily CBD oil ingestion.

We expect that CBD-treated patients will show equivalent levels of side effects as those receiving placebo oil.

STUDY METHODS AND PROCEDURES

Participant Recruitment: 150 participants between the ages of 18 and older will be recruited through several outlets including notices posted on campus, announcements on our research laboratory website and national organizations related to PTSD and its treatment.

Participant Screening: Participants will undergo a two-stage screening procedure. Stage 1 will be a brief structured web-based screening interview. Stage 2 will be a web-based, self-report version of the Mini-International Neuropsychiatric Interview (MINI). Participants meeting the following inclusion and exclusion enrollment criteria will be invited to take part in the study (see below).

NOTE: ALL STUDY PROCEDURES ARE COMPLETED AT PARTICIPANTS' HOMES. NO VISITS TO OUR RESEARCH LABORATORY ARE REQUIRED.

Inclusion/Exclusion Criteria:

1. Meets for a current DSM-5 diagnosis of PTSD as their "primary" mental disorder
2. Age between 18+
3. Fluent in English
4. Willingness to provide signed informed consent online
5. No history of a suicide attempt in the past 6 months
6. No history of psychosis within the past 6 months

9. No history of current alcohol or substance use disorder within the past month.

10. No current medical problems that would preclude safe ingestion of CBD oil 11. Willingness to refrain from other forms of Cannabis use during the study period 12. Has home access to the internet. 13. No history of adverse reaction to CBD. 14. No allergy to coconut oil.

Participant Informed Consent:

All study participants will be consented by the study coordinator or a doctoral student research assistant. The online informed consent document will provide participants with information regarding the aims of the project, what they will be asked to do, any anticipated risks or benefits associated with participating in the study, as well as a clear statement that their participation is voluntary and that they may discontinue participation at any time.

Study Design Overview: The research plan is to conduct a Phase II double-blind placebo controlled randomized clinical trial comparing the efficacy of two CBD oil formulations (CBD Isolate (300 mg/day) and CBD Broad Spectrum versus Placebo Oil.

CBD/Placebo Dosing:

Nightly dosing of a hemp-derived formulation of purified CBD isolate (300 mg), CBD Broad Spectrum (300 mg.) or matching placebo oil daily for 8 weeks. Individual doses of both CBD formulations and placebo oil will be provided in identical individual plastic syringes. All patients, PI, and staff who interact with study participants will be blind to participants' assigned treatment condition.

Clinical Assessment Schedule:

Week 0 - Pre-Treatment Screening Visit: All enrolled study participants will complete from their home a clinical assessment battery consisting of self-report rating scales over the Internet (see measures).

Treatment Visits (Weeks 1 - 8): During this phase, all study participants will (a) receive via USPS their weekly allotment of CBD/Placebo oil; (b) complete weekly clinical status assessments via the Internet (see measures).

Posttreatment Assessment Visit (Week 9): All participants will complete an online battery of clinical outcome measures identical to those administered during their pre-treatment visit (see outcome measures).

1-Month Follow-up Assessment Visit (Week 13): All participants will be re-administered the complete battery of primary and secondary outcome measures (see outcome measures).

Outcome Measures

Primary Clinical Outcomes: The primary clinical outcome will be scores on the PTSD Checklist for DSM-5 (PCL-5). Models will be coded to test differences between (1) CBD Isolate + Broad Spectrum vs. Placebo and (2) CBD Isolate vs CBD Broad Spectrum at the primary endpoint (post-treatment) and secondary endpoint (1-month follow-up).

Secondary Clinical Outcomes: Several additional psychiatric outcomes will be assessed at post treatment and follow-up. These clinical outcomes and their respective measures appear below.

* Depression (PHQ-9)
* Disability (SDS)
* Quality of Life (WHOQOL-BREF)
* Anxiety (GAD-7)
* Alcohol Use (PROMIS Alcohol Use -Short Form).

Data Management Data Management involves development of methods for ensuring that data collection instruments are programmed; data are properly collected; participants are tracked and monitored over the course of the study; data sets are documented and maintained; variables are created and documented; and main analyses are conducted. To enhance quality control, all data for the current study including demographic information, diagnoses, and participant and clinician rated measures will be directly entered into a HIPAA-compliant electronic case report form (eCRF) using Qualtrics - a secure cloud-based platform designed exclusively for supporting HIPAA compliant data capture and storage. Qualtrics provides: (a) An intuitive interface for data entry with data validation; (b) Audit trails for tracking data manipulation and export procedures; (c) Procedures for importing data from external sources; (d) Automated export procedures for seamless data downloads to common statistical packages (SPSS, SAS, Stata, R) to facilitate data analysis; (e) automated and secure data back-up and storage to servers housed at the University of Texas Population Research Center (PRC). Dr. Telch in his role as Principal Investigator will serve as the Senior data manager and will meet bi-weekly with the research staff on issues related to data management.

ELIGIBILITY:
Inclusion Criteria:

1. Meets for a current DSM-5 diagnosis of PTSD as their "primary" mental disorder
2. Age 18 or older
3. Fluent in English
4. Has access to the internet
5. Willingness to provide signed informed consent
6. Willingness to refrain from all non-study cannabis use during the study period

Exclusion Criteria:

1. History of a suicide attempt within the past 6 months
2. History of psychosis within the past 6 months
3. History of current alcohol or substance use disorder within the past month
4. Any medical problems that would preclude participating in the study
5. History of adverse reaction to CBD oil or other CBD products
6. Allergy to coconut oil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
PCL-5 | Post-treatment (week 9) and one month (week 13) follow-up assessments
  Change from baseline in patient-rated symptoms of PTSD.

SECONDARY OUTCOMES:
PHQ-9 | Post-treatment (week 9) and one month (week 13) follow-up assessments
  Change from baseline in patient-rated symptoms of depression.
SDS | Post-treatment (week 9) and one month (week 13) follow-up assessments
  Change from baseline in overall disability.
WHOQOL-BREF | Post-treatment (week 9) and one month (week 13) follow-up assessments
  Change from baseline in quality of life.
GAD-7 | Post-treatment (week 9) and one month (week 13) follow-up assessments
  Change from baseline in patient-rated symptoms of anxiety.
PROMIS Alcohol Use -Short Form | Post-treatment (week 9) and one month (week 13) follow-up assessments
  Change from baseline in patient-rated alcohol use.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Telch, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- Laboratory for the Study of Anxiety Disorders, University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shalev AY, Gevonden M, Ratanatharathorn A, Laska E, van der Mei WF, Qi W, Lowe S, Lai BS, Bryant RA, Delahanty D, Matsuoka YJ, Olff M, Schnyder U, Seedat S, deRoon-Cassini TA, Kessler RC, Koenen KC; International Consortium to Predict PTSD. Estimating the risk of PTSD in recent trauma survivors: results of the International Consortium to Predict PTSD (ICPP). World Psychiatry. 2019 Feb;18(1):77-87. doi: 10.1002/wps.20608. PMID 30600620
- [Background] Powers MB, Gillihan SJ, Rosenfield D, Jerud AB, Foa EB. Reliability and validity of the PDS and PSS-I among participants with PTSD and alcohol dependence. J Anxiety Disord. 2012 Jun;26(5):617-23. doi: 10.1016/j.janxdis.2012.02.013. Epub 2012 Mar 3. PMID 22480715
- [Background] Merikangas KR, Akiskal HS, Angst J, Greenberg PE, Hirschfeld RM, Petukhova M, Kessler RC. Lifetime and 12-month prevalence of bipolar spectrum disorder in the National Comorbidity Survey replication. Arch Gen Psychiatry. 2007 May;64(5):543-52. doi: 10.1001/archpsyc.64.5.543. PMID 17485606
- [Background] Powers MB, Halpern JM, Ferenschak MP, Gillihan SJ, Foa EB. A meta-analytic review of prolonged exposure for posttraumatic stress disorder. Clin Psychol Rev. 2010 Aug;30(6):635-41. doi: 10.1016/j.cpr.2010.04.007. Epub 2010 May 2. PMID 20546985
- [Background] White CM. A Review of Human Studies Assessing Cannabidiol's (CBD) Therapeutic Actions and Potential. J Clin Pharmacol. 2019 Jul;59(7):923-934. doi: 10.1002/jcph.1387. Epub 2019 Feb 7. PMID 30730563
- [Background] Devinsky O, Cross JH, Laux L, Marsh E, Miller I, Nabbout R, Scheffer IE, Thiele EA, Wright S; Cannabidiol in Dravet Syndrome Study Group. Trial of Cannabidiol for Drug-Resistant Seizures in the Dravet Syndrome. N Engl J Med. 2017 May 25;376(21):2011-2020. doi: 10.1056/NEJMoa1611618. PMID 28538134
- [Background] Devinsky O, Patel AD, Cross JH, Villanueva V, Wirrell EC, Privitera M, Greenwood SM, Roberts C, Checketts D, VanLandingham KE, Zuberi SM; GWPCARE3 Study Group. Effect of Cannabidiol on Drop Seizures in the Lennox-Gastaut Syndrome. N Engl J Med. 2018 May 17;378(20):1888-1897. doi: 10.1056/NEJMoa1714631. PMID 29768152
- [Background] McGuire P, Robson P, Cubala WJ, Vasile D, Morrison PD, Barron R, Taylor A, Wright S. Cannabidiol (CBD) as an Adjunctive Therapy in Schizophrenia: A Multicenter Randomized Controlled Trial. Am J Psychiatry. 2018 Mar 1;175(3):225-231. doi: 10.1176/appi.ajp.2017.17030325. Epub 2017 Dec 15. PMID 29241357
- [Background] Bergamaschi MM, Queiroz RH, Chagas MH, de Oliveira DC, De Martinis BS, Kapczinski F, Quevedo J, Roesler R, Schroder N, Nardi AE, Martin-Santos R, Hallak JE, Zuardi AW, Crippa JA. Cannabidiol reduces the anxiety induced by simulated public speaking in treatment-naive social phobia patients. Neuropsychopharmacology. 2011 May;36(6):1219-26. doi: 10.1038/npp.2011.6. Epub 2011 Feb 9. PMID 21307846
- [Background] Berk M, Ng F, Dodd S, Callaly T, Campbell S, Bernardo M, Trauer T. The validity of the CGI severity and improvement scales as measures of clinical effectiveness suitable for routine clinical use. J Eval Clin Pract. 2008 Dec;14(6):979-83. doi: 10.1111/j.1365-2753.2007.00921.x. Epub 2008 May 2. PMID 18462279
- [Background] Pinto-Meza A, Serrano-Blanco A, Penarrubia MT, Blanco E, Haro JM. Assessing depression in primary care with the PHQ-9: can it be carried out over the telephone? J Gen Intern Med. 2005 Aug;20(8):738-42. doi: 10.1111/j.1525-1497.2005.0144.x. PMID 16050884
- [Background] Leon AC, Olfson M, Portera L, Farber L, Sheehan DV. Assessing psychiatric impairment in primary care with the Sheehan Disability Scale. Int J Psychiatry Med. 1997;27(2):93-105. doi: 10.2190/T8EM-C8YH-373N-1UWD. PMID 9565717
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Derived] Telch MJ, Fischer CM, Zaizar ED, Rubin M, Papini S. Use of Cannabidiol (CBD) oil in the treatment of PTSD: Study design and rationale for a placebo-controlled randomized clinical trial. Contemp Clin Trials. 2022 Nov;122:106933. doi: 10.1016/j.cct.2022.106933. Epub 2022 Sep 22. PMID 36154908